CLINICAL TRIAL: NCT06301724
Title: A Randomized Double-blind Trial to Explore Effectiveness of Stellate Ganglion Block in Individuals With Parkinson's Disease
Brief Title: Effectiveness of Stellate Ganglion Block in Individuals With Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-PKS
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Injections; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block (Experimental): the patients were provided with stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g)
  Interventions: Procedure: Injection; Drug: Lidocaine hydrochloride
- Injection (Placebo Comparator): the patients were provided with injection, which was with the same procedure of stellate ganglion block but no drugs.
  Interventions: Procedure: Injection

INTERVENTIONS:
Procedure: Injection — The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
Drug: Lidocaine hydrochloride — the patients were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: Lidocaine
  Arms: Stellate ganglion block

SUMMARY:
The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia and activities of daily living in patients with Parkinson's disease.

Participants will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

DETAILED DESCRIPTION:
Dysphagia, or swallowing difficulty, is a common symptom associated with Parkinson's disease. It is characterized by weakened chewing and throat muscles, leading to difficulties in eating, coughing, and a sensation of choking in individuals with Parkinson's disease.

The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia and activities of daily living in patients with Parkinson's disease.

Participants will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the - - Chinese Medical Association in 2006.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 10
  Penetration-Aspiration Scale is used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food enter the airway and caused penetration or aspiration during the swallowing process. As the level increases, the severity of dysphagia also increases.The scores rang from 0 to 8

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 10
  activities of daily living of patients will be assessed using the modified Barthel Index . The scale includes 10 items such as feeding, bathing, walking, dressing. Each item is rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There is a positive correlation between activities of daily living and the final score.
Functional Oral Intake Scale | day 1 and day 10
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No